CLINICAL TRIAL: NCT07176351
Title: Acceptability and Feasibility of Extended-Release Subcutaneous Buprenorphine on a Mobile Pharmacy Clinic: A Pilot Study
Brief Title: Acceptability and Feasibility of Extended-Release Subcutaneous Buprenorphine on a Mobile Pharmacy Clinic
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Braeburn Inc (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2000040545
Record Dates: First submitted 2025-09-08; First posted 2025-09-16 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Opioid Use Disorder
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Buprenorphine

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Buprenorphine (Experimental): Participants will be offered weekly or monthly Buprenorphine injections
  Interventions: Drug: Buprenorphine

INTERVENTIONS:
Drug: Buprenorphine — Weekly or monthly extended-release subcutaneous injection
  Other Names: BRIXADI

SUMMARY:
This exploratory project will assess the acceptability and feasibility of monthly extended-release subcutaneous buprenorphine (BRIXADI; XR-B) to treat opioid use disorder (OUD) among persons in the community receiving care on a mobile pharmacy clinic (MPC).

Participants who are interested in initiating monthly or weekly injections of subcutaneous XR-B (BRIXADI) as a treatment for their OUD will be enrolled in a 6-month study assessing the acceptability and feasibility of receiving XR-B on an MPC.

DETAILED DESCRIPTION:
This is a prospective cohort study, participants will be able to have a shared decision with the clinician if they would like to receive XR-B. The medication would be available for free for 6 months to determine the acceptability and feasibility of being able to provide XR-B from the first mobile pharmacy clinic in the nation. Medical visit data will be collected for 6 months along with medical record data.

BRIXADI (by Braeburn), subcutaneous long-acting buprenorphine in weekly and monthly formulations will be used for this project. Participants will be engaged in shared decision making with a project clinician regarding the weekly or monthly formulation. Dosing will be based on medical need. Participants will be able to access to free medication for 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Able to provide written informed consent in English or Spanish
* Current or history of DSM-5 moderate-to-severe OUD per Rapid Opioid Use Disorder Assessment (ROUDA)
* Not planning to move out of state or to new location during study enrollment.

Exclusion Criteria:

* Medical or psychiatric disorders making participation unsafe or regular follow-up unlikely, (such as suicidal ideation or pre-existing moderate to severe hepatic impairment)
* Persons who are pregnancy
* People who show violent or threatening behavior toward staff and/or others
* Allergy, hypersensitivity, or medical contraindication to medication (the BRIXADI needle cap is synthetically derived from natural rubber latex which may cause allergic reactions in persons with latex-sensitivity)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2027-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Retention of XR-B at month 6 | Month 6
  Proportion of participants that were retained on 6 months of XR-B injections.

CONTACTS AND LOCATIONS:
Overall Officials: Sandra Springer, MD, Principal Investigator — Yale University
Locations (1):
- Yale School of Medicine, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No